CLINICAL TRIAL: NCT06196632
Title: Development and Validation of Logistic Regression Models to Predict Durable Functional Cure in Patients With Chronic Hepatitis B After Pegylated Interferon Alpha-2b Based Therapy
Brief Title: Development and Validation of Models to Predict Functional Cure in Patients With CHB After Peg-IFN Based Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-2023(ZM)-726
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-12

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Nucleosides

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- "de novo" strategy-HBeAg positive: HBeAg positive patients treated with simultaneous administration of NA and Peg-IFN
  Interventions: Drug: Peginterferon-α; Nucleoside analogs
- "de novo" strategy-HBeAg negative: HBeAg positive patients treated with simultaneous administration of NA and Peg-IFN
  Interventions: Drug: Peginterferon-α; Nucleoside analogs
- "add-on" strategy-HBeAg positive: HBeAg positive patients treated with NA followed by addition of Peg-IFN.
  Interventions: Drug: Peginterferon-α; Nucleoside analogs
- "add-on" strategy-HBeAg negative: HBeAg negative patients treated with NA followed by addition of Peg-IFN.
  Interventions: Drug: Peginterferon-α; Nucleoside analogs

INTERVENTIONS:
Drug: Peginterferon-α; Nucleoside analogs — Patients with chronic hepatitis B were treated with the combination of peginterferon-α and nucleoside analogs

SUMMARY:
Hepatitis B virus (HBV) infection is prevalent across the world. Functional cure is the optimal endpoint of antiviral therapy for chronic hepatitis B virus (HBV) infection. Currently available anti-HBV therapy includes nucleoside analogs (NAs) and peginterferon-α (Peg-IFNα). Combination of Peg-IFNα and NAs, each with different mechanisms of action, is an attractive approach for treating chronic HBV infection. In this study, we aim to establish logistic regression models to predict durable functional cure in patients with CHB treated by combination of Peg-IFNα and NAs, which might be useful for clinical physicians to make personalized treatment decisions. These models will be constructed using baseline routine clinical laboratory indicators with high diagnostic accuracy. These models might be widely applicable to almost all medical institutions and will effectively promote the application of Peg IFN α plus NAs therapy in clinical work. The findings in this study might greatly improve the functional cure rate of CHB and reducing the incidence rate and mortality of HBV related end-stage liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign an informed consent form;
* 2. HBsAg (+), and the course of the disease exceeds six months;
* 3. Age range from 16 to 70 years old;
* 4. Female participants of childbearing age who had a negative pregnancy test before the trial and were able to take effective contraceptive measures;
* 5. During the treatment period, within six months after the end of treatment, the patients agrees to use contraception

Exclusion Criteria:

* 1. Patients with a known history of allergy to Peg-IFNα and NAs;
* 2. Co-infection with other virus such as HAV, HCV, HDV, HEV, HIV, etc;
* 3. Patients with liver cirrhosis or a Child Pugh score of 7 or above;
* 4. History or evidence of liver disease caused by other factors (such as autoimmune liver disease, alcoholic liver disease, non-alcoholic fatty liver disease, drug-induced hepatitis, hepatolenticular degeneration, etc.);
* 5. Pregnant or lactating women; Have a history of alcohol or drug abuse within the year prior to the trial enrollment screening;
* 6. Neutrophil count<1.5 × 109/L or hemoglobin<100g/L or platelet count<80 × 109/L; During the trial enrollment screening, serum creatinine was higher than the upper normal limit;
* 7. A history of severe diseases in important organs and tissues such as the heart, brain, kidneys, retina, and muscles;
* 8. Having a history of mental illness or a family history of mental illness, or a Hamilton Depression Scale score greater than 7 points;
* 9. History of endocrine system or autoimmune diseases, such as thyroid disease, diabetes, systemic lupus erythematosus, sarcoidosis, autoimmune thrombocytopenic purpura, etc;
* 10. History of malignant tumors;
* 11. During the trial enrollment screening, suspicious liver malignant tumors were detected by ultrasound, or AFP was greater than 100ng/mL or AFP cannot remain stable within 3 months prior to the experiment;
* 12. Has a history of important organ transplantation;
* 13. Other diseases that researchers believe are not suitable for inclusion.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants were retrospectively enrolled from more than 10 hospitals in China.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-06 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional cure of chronic hepatit B | 48 weeks
  The level of hepatitis B surface antigen (HBsAg) is below 0.05IU/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Liu HH, Jiang XM, Cui C, Zhao J, Xu J, Wang SK, Hu LH, Yin YP, Wang X, Yu LJ, Xu C, Zhao ZH, Xing YQ, Liu Y, Wang K, Gao S. Development and Validation of a Predictive Model for HBsAg Seroclearance After Peg-IFN-Based Therapy: A Multicentre Study. Drug Des Devel Ther. 2025 Nov 7;19:9973-9982. doi: 10.2147/DDDT.S545700. eCollection 2025. PMID 41229921